CLINICAL TRIAL: NCT06203691
Title: Nirvana Super Pro Supplementation in Orthopedic Surgery Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nirvana Water Sciences Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11495
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Arthropathy of Knee; Arthropathy of Hip
Keywords: Arthroplasties; Knee & Hip Replacement; Dietary Supplements
MeSH Terms: interventions — Dietary Supplements; Control Groups

STUDY DESIGN:
Intervention Model Description: One group will receive the supplements. The control group will not receive the supplements. All participants will undergo strength test - pre and post operatively.
Who Masked: Care Provider
Masking Description: Participants will be assigned a number and by the care provider staff prior to providing collecting data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement Group (Experimental): 50 of the 100 participants will be given supplements (Prepare & Recover) for pre & post operation.
  Interventions: Dietary Supplement: Supplementation with Nirvana Super Pro Liquid Supplements
- Non-Supplement Group (Placebo Comparator): No supplements will be given to the non-supplement group.
  Interventions: Dietary Supplement: Non-Supplementation Group

INTERVENTIONS:
Dietary Supplement: Supplementation with Nirvana Super Pro Liquid Supplements — Intervention will measure strength pre & post operatively. Intervention group will receive liquid supplements (3oz daily shots) pre (Prepare) and Post (Recover) operatively.
  Arms: Supplement Group
Dietary Supplement: Non-Supplementation Group — Intervention will measure strength pre & post operatively. Intervention group will not receive liquid supplements.
  Other Names: Control Group
  Arms: Non-Supplement Group

SUMMARY:
The purpose of this study is to investigate orthopedic patients undergoing either a total hip replacement (THR) or total knee arthroplasty (TKR) using two dietary supplements, PREPARE and RECOVER, and their recovery times post-surgery.

DETAILED DESCRIPTION:
This study involves two dietary supplements that have been formulated by Nirvana Water Sciences Corp for Super Inspired LLC. A pre-operative supplement, called PREPARE, has been created with HMB, Vitamin D, Selenium, Zinc, and Vitamin C to provide pre-operative nutrition, promote lean muscle development and boost immunity. A post-operative supplement, called RECOVER, has been created with HMB, collagen, L-citrulline, resveratrol, and 2-HOBA to help maintain lean muscle, support wound healing and reduce oxidative stress.

HMB or βeta-hydroxy βeta-methylbutyrate is a nutritional supplement that has been extensively studied for its potential benefits. It is a substance that your body naturally produces when it breaks down the amino acid leucine, which is essential for protein synthesis and muscle repair. There are over 50 human studies, 40 review articles and four meta-analyses showing its effectiveness and safety. These clinical studies provide evidence of the benefits of HMB and supports the claims that HMB boosts muscle performance, slows muscle degradation, and reduces muscle recovery time.

Muscle atrophy (loss of muscle mass) and poor muscle function are demonstrated in patients suffering from osteoarthritis (OA) involving several joints and particularly the hip and the knee joints. Several studies have shown that this atrophy is worsened in the immediate postoperative period, and complete recovery is not established up to 2 years postop. Little is known about muscular recovery after either total hip replacement (THR) or total knee arthroplasty (TKR).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects will be enrolled into the study.
* Age ≥45-80 years.
* Free of liver and kidney diseases, and with no evidence of uncontrolled hypertension.
* Does not have a chronic disease that affects calcium or bone metabolism (i.e., asthma with chronic use of high dose steroids, inflammatory bowel disease, Crohn's disease, primary hyperparathyroidism, seizure disorder with use of phenobarbital, etc.).
* Not classified as morbidly obese (body mass index (BMI) >43 kg/m2).
* Six weeks since major surgery (three weeks since minor surgery).
* Total joint replacement is not a revision of previous joint replacement.
* Willing to consume dietary supplements for the study period.
* Individuals diagnosed with osteoporosis, or a bone density >2.0 standard deviations below the mean, will not be enrolled in the study.
* No other serious medical illness.
* Physicians have placed no restriction on physical exercise.
* Patient is scheduled for a total knee or hip replacement and agrees to consume the 28-day pre-operative regime.

Exclusion Criteria:

* Evidence of liver and kidney diseases, uncontrolled hypertension, or Type I or II diabetes mellitus requiring insulin for glucose control.
* The presence of a chronic disease that affects calcium or bone metabolism (i.e., asthma with chronic use of high dose steroids, inflammatory bowel disease, Crohn's disease, primary hyperparathyroidism, seizure disorder with use of phenobarbital, etc.).
* Classified as morbidly obese (body mass index (BMI) >43 kg/m2).
* Less than six weeks since major surgery or three weeks since minor surgery.
* Surgery is a revision of a previous total joint replacement.
* Not willing to consume nutritional supplements for the study period.
* Individuals diagnosed with osteoporosis, or a bone density >2.0 standard deviations below the mean, will not be enrolled in the study.
* Other serious medical illness, which the subject's doctor or medical review team has decided affects the subject's ability to participate in the study. For example, pathological hip fracture or cancer disease in active phase or undergoing treatment (radiotherapy or chemotherapy).
* History of blood clots and/or the use of blood thinning medications
* Subjects on high dose vitamin D therapies (i.e., 50,000 IU vitamin D).

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 30+ days prior to surgery, 14-days after surgery, 28-30 days after surgery
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a questionnaire that measures the impact of osteoarthritis on pain, stiffness, and physical function in the hip or knee joints. It is a self-administered tool that consists of 24 items, each rated on a scale of 0 to 4, with higher scores indicating worse symptoms. The WOMAC is widely used in clinical trials and research studies to evaluate the effectiveness of treatments and interventions for osteoarthritis.
Timed Up & Go (TUG) | 30+ days prior to surgery, 14-days after surgery, 28-30 days after surgery
  The Timed Up and Go test or TUG test is used to help evaluate mobility. It is a simple test that measures how quickly one can stand up, walk 10 feet, turn around, walk back, and sit down. It is often done to assess mobility in older adults or predict their risk of falls.
Grip Strength using a Jamar Hydraulic Hand Dynamometerer | 30+ days prior to surgery, 14-days after surgery, 28-30 days after surgery
  Grip Strength is a measure of the maximum force or tension generated by one's forearm muscles when gripping an object. A Jamar Hydraulic Hand Dynamometer is a device that can measure this force in pounds or kilograms. It is commonly used by physical therapists, occupational therapists, and hand surgeons to assess grip strength and monitor recovery or rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Candice St. Pierre, Ph.D., Study Chair — Nirvana Water Sciences Corp
Locations (1):
- University Orthopedics Center, Altoona, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Masked IDP data will be shared with researchers for statistical analysis and conclusions.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available for 2 months for statistical analysis.
Access Criteria: Data will be securely shared and only masked participant data will be shared with researchers.

REFERENCES:
- [Background] Bear DE, Langan A, Dimidi E, Wandrag L, Harridge SDR, Hart N, Connolly B, Whelan K. beta-Hydroxy-beta-methylbutyrate and its impact on skeletal muscle mass and physical function in clinical practice: a systematic review and meta-analysis. Am J Clin Nutr. 2019 Apr 1;109(4):1119-1132. doi: 10.1093/ajcn/nqy373. PMID 30982854
- [Background] Hiemstra LA, Gofton WT, Kriellaars DJ. Hip strength following hamstring tendon anterior cruciate ligament reconstruction. Clin J Sport Med. 2005 May;15(3):180-2. doi: 10.1097/01.jsm.0000157795.93004.ea. PMID 15867563
- [Background] Nishizaki K, Ikegami H, Tanaka Y, Imai R, Matsumura H. Effects of supplementation with a combination of beta-hydroxy-beta-methyl butyrate, L-arginine, and L-glutamine on postoperative recovery of quadriceps muscle strength after total knee arthroplasty. Asia Pac J Clin Nutr. 2015;24(3):412-20. doi: 10.6133/apjcn.2015.24.3.01. PMID 26420181
- [Background] Silva AM, Shen W, Heo M, Gallagher D, Wang Z, Sardinha LB, Heymsfield SB. Ethnicity-related skeletal muscle differences across the lifespan. Am J Hum Biol. 2010 Jan-Feb;22(1):76-82. doi: 10.1002/ajhb.20956. PMID 19533617
- [Background] Wilkinson DJ, Hossain T, Hill DS, Phillips BE, Crossland H, Williams J, Loughna P, Churchward-Venne TA, Breen L, Phillips SM, Etheridge T, Rathmacher JA, Smith K, Szewczyk NJ, Atherton PJ. Effects of leucine and its metabolite beta-hydroxy-beta-methylbutyrate on human skeletal muscle protein metabolism. J Physiol. 2013 Jun 1;591(11):2911-23. doi: 10.1113/jphysiol.2013.253203. Epub 2013 Apr 3. PMID 23551944
- [Background] Wu H, Xia Y, Jiang J, Du H, Guo X, Liu X, Li C, Huang G, Niu K. Effect of beta-hydroxy-beta-methylbutyrate supplementation on muscle loss in older adults: a systematic review and meta-analysis. Arch Gerontol Geriatr. 2015 Sep-Oct;61(2):168-75. doi: 10.1016/j.archger.2015.06.020. Epub 2015 Jul 3. PMID 26169182